Status

# POST-MARKETING OBSERVATIONAL STUDY PROTOCOL HUM04-28

A five-year, post-marketing observational study to follow-up patients with rheumatoid arthritis, psoriatic arthritis or ankylosing spondylitis who are treated with HUMIRA® (adalimumab)

Date

Version

| 1.0 | 26 November 2018 | Final |
|------------|------------------|-------|
| Approvals | | |
| Signature: | Date: | |
| Signature: | Date: | _0 |

# TABLE OF CONTENTS

| 1. M | ETHODOLOGY | .3 |
|------|----------------------|-----|
| | Study Objective | |
| | AVAILABLE DATA | |
| | PATIENT POPULATION | |
| 1.4 | Data Handling | . 3 |
| 1.5 | DERIVED DATA | . 4 |
| 2 | STATISTICAL ANALYSIS | 5 |

#### 1. METHODOLOGY

The purpose of this statistical analysis plan is to provide detailed information on the statistical analysis of the data of the ProAct study. The plan is based on the quotation dated 18 October 2017 and the mail dated 4 April 2017.

### 1.1 Study Objective

To evaluate the effectiveness and safety of adalimumab for the treatment of rheumatoid arthritis (RA), psoriatic arthritis (PsA) and ankylosing spondylitis (AS) in real life clinical practice.

#### 1.2 Available data

The questionnaires table, as received on 5 February 2018, contained 47378 records, of which 5947 baseline visits. This database has been adapted by hardcoding in the programmation in order to resolve inconsistencies, double patients, misclassification of visits, add additional visit CRF pages, add additional AE pages. A total of 5920 patients of which 2836 rheumatoid arthritis patients, 1127 psoriatic arthritis patients (of which 197 Oligoarticular PsA) and 1957 ankylosing spondylitis patients were included in the analysis.

The parameter DAS28 was entered in the database from the moment the new Belgium reimbursement criteria for Humira were in place (2010).

Visits were scheduled at baseline, months 3, 6, 9 and 12, then every 6 months till 5 years.

## 1.3 Patient Population

All patients are to be considered in the analysis.

## 1.4 Data Handling

All data handling rules used during the analysis will be described in the section Methodology of the Statistical Report.

'LT' visits are visits added in the database for patients who were lost to follow-up in order to close the patient in the database. These visits will not be taken into account for any analysis.

#### 1.5 Derived Data

- Study duration (year) = (visit date of last visit visit date of baseline visit)/365.25
- Completed patients: patients with >= 1734 days study duration
- Treatment duration (year):

For completed patients:

(Date of last visit – Date of baseline visit)/365.25

For not completed patients:

Sum of number of weeks/52, months/12 and years patient has been on drug documented on the last visit

If missing: (Date of last visit – Date of baseline visit)/365.25

Note: Some patients stopped Humira temporaly. The periods of not taken Humira are not taken into account for the analysis. These patients will be considered as having taken Humira during the complete study.

- Treatment duration category:
  - 0 to 3 months
  - > 3 to 6 months
  - > 6 to 9 months
  - > 9 to 12 months
  - > 12 to 18 months
  - > 18 to 24 months
  - > 24 to 30 months
  - > 30 to 36 months
  - > 36 to 42 months
  - > 42 to 48 months
  - > 48 to 54 months > 54 to 60 months
  - > 60 months
- For the purpose of the analysis of the evolution of parameters over time, follow-up visits will be classified into time windows, defined upon the number of days between Visit 1 and the date of each subsequent visit (PERIOD = Date of follow-up visit Date of Visit 1)
  - Period = Date of visit Date of baseline visit
  - Month 3 window: 1 <= period <= 137 days
  - Month 6 window: 138 <= period <= 228 days
  - Month 9 window: 229 <= period <= 319 days
  - Month 12 window: 320 <= period <= 456 days
  - Month 18 window: 457 <= period <= 639 days
  - Month 24 window: 640 <= period <= 821 days
  - Month 30 window: 822 <= period <= 1004 days

- Month 36 window: 1005 <= period <= 1186 days
- Month 42 window: 1187 <= period <= 1368 days
- Month 48 window: 1369 <= period <= 1551 days
- Month 54 window: 1552 <= period <= 1733 days
- Month 60 window: 1734 <= period <= 1916 days

Each visit will be classified in a time window. If the date of the visit is completely missing, it will be assumed that the visit took place on the target day of the window as indicated on top of the follow-up page. If more than one follow-up visit is classified into the same time window, the visit closest to the target day is retained. If within a time window there are two visits at the same distance from the target day, the visit which comes first (e.g. before the target date) is retained. If there are two visits on the same date, the first record is retained.

- BASDAI responder: a relative improvement in BASDAI of >= 50%
- DAS28 category:  $<2.6, \ge 2.6$  and  $\le 3.2, >3.2$
- Serious adverse event = event where at least one criteria of seriousness is present
- An adverse event is considered to start in a certain year if the difference between start date and date of baseline (=AEPER) is in the following windows:
  - Year 1:  $0 \le AEPER \le 365.25$
  - Year 2:  $365.25 \le AEPER < 730.5$
  - Year 3 730.5 <= AEPER < 1095.75
  - Year 4: 1095.75 <= AEPER < 1461
  - Year 5: 1461 <= AEPER < 1826.25

#### 2 STATISTICAL ANALYSIS

The analysis of the baseline data and prior anti-TNF treatment will be performed broken down by indication (RA, PsA, AS). Within each indication, baseline data will also presented broken down by completed/not completed patients. Statistical tests will be performed to compare baseline data for patients completed/not completed the study.

The analysis of treatment duration and the evolution of different parameters over time, will be performed broken down by indication (RA, PsA, AS).

The analysis of adverse events will be performed for all patients together and broken down by indication (RA, PsA, AS):

- Overall
- Per year (up to 5 years)
- By cumulative yearly period (till 5 years)
- Incidence
- Incidence divided by total exposure to treatment (till 5 years).
- Reason for seriousness
- Serious adverse events: number of patients and incidence by system organ class and preferred term
- Non-serious adverse events: number of patients by system organ class and preferred term

If an adverse event has no onset date, the observation date will be taken as onset date. Events that are coded with multiple MedDRA Terms will be counted as separate event.

The percentages in the adverse event table are calculated as follows:

| Table | Nominator | Denominator |
|---|---|---|
| Number of patients with an | Number of patients treated | Number of patients treated |
| adverse event per year. | in that year with at least one | in that year. |
| | adverse event in that year. | |
| Number of patients with an | Number of patients with at | Number of patients. |
| adverse event per | least one adverse event in | _ |
| cumulative year | that year or before. | |
| Number of adverse events | Number of adverse events in | The sum of the patients' |
| by total exposure to | that year or before. | treatment exposure time in |
| treatment | | that year or before. |

The following tables will be presented:

# **Rheumatoid Arthritis**

| 1 | Baseline Characteristics – All Patients and Broken Down by Early Termination |
|---|---|
| 1.1 | Age |
| 1.2 | Gender |
| 1.3 | Disease Duration Before Inclusion |
| 1.4 | Anti-TNF use Before Inclusion |
| 1.4.1 | Anti-TNF Naïve / Experienced |
| 1.4.2 | Types of Anti-TNF use Before Inclusion |
| 1.5 | Physician's Assessment of Disease Activity |
| 1.6 | Clinical Examination |
| 1.6.1 | Joint Assessment (tender joints count, swollen joints count) |
| 1.6.2 | Inflammatory Parameters (CRP, ESR) |
| 1.6.3 | Physical Function (HAQ %) |
| 1.7 | Concomitant Medication |
| 1.7.1 | Concomitant Steroids |
| 1.7.2 | Concomitant NSAIDs |
| 1.7.3 | Concomitant Immunomodulators |
| 1.7.4 | Number of DMARDs Used |
| 1.7.5 | Frequency of Use of Each Type of DMARD |
| 1.7.6 | Combination of Types of DMARD Used |
| 1.8 | Study Duration |
| 1.9 | Results of the Tests |
| _ | E-II D-4- |
| 2 | Follow-up Data |
| 2<br>2.1 | Treatment Duration |
| | <u>-</u> |
| 2.1 | Treatment Duration |
| 2.1<br>2.1.1 | Treatment Duration Treatment Duration |
| 2.1<br>2.1.1<br>2.1.2 | Treatment Duration Treatment Duration Treatment Duration Category |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) in Each Window Physical Function (HAQ %) - Difference from Baseline Physical Function (HAQ %) - Number of Patients with >7.33% Reduction from |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5<br>2.3.6 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) in Each Window Physical Function (HAQ %) - Difference from Baseline Physical Function (HAQ %) - Number of Patients with >7.33% Reduction from Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5<br>2.3.6<br>2.3.7 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) in Each Window Physical Function (HAQ %) - Difference from Baseline Physical Function (HAQ %) - Number of Patients with >7.33% Reduction from Baseline DAS28 in Each Window |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5<br>2.3.6<br>2.3.7 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) in Each Window Physical Function (HAQ %) - Difference from Baseline Physical Function (HAQ %) - Number of Patients with >7.33% Reduction from Baseline |

| 3 | Adverse Events |
|---|---|
| 3.1 | Adverse Events |
| 3.1.1 | Patients with Adverse Events, Patients with Serious Adverse Events, Patients with Fatal Adverse Events and Patients with Adverse Events Causing Treatment Discontinuation |
| 3.1.2 | Patients with Adverse Events by MedDRA System Organ Class |
| 3.1.3 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.2 | Adverse Events per Year |
| 3.2.1 | Patients with Adverse Events, Patients with Serious Adverse Events, Patients with Fatal Adverse Events and Patients with Adverse Events Causing Treatment Discontinuation |
| 3.2.2 | Patients with Adverse Events by MedDRA System Organ Class |
| 3.2.3 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.3 | Adverse Events by Cumulative Yearly Period |
| 3.3.1 | Patients with Adverse Events, Patients with Serious Adverse Events, Patients with Fatal Adverse Events and Patients with Adverse Events Causing Treatment Discontinuation |
| 3.3.2 | Patients with Adverse Events by MedDRA System Organ Class |
| 3.3.3 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.4 | Incidence Adverse Events |
| 3.4.1 | Number of Adverse Events, Serious Adverse Events, Fatal Adverse Events and Number of Adverse Events Causing Treatment Discontinuation |
| 3.4.2 | Number of Adverse Events by MedDRA System Organ Class |
| 3.4.3 | Number of Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.5 | Incidence Adverse Events Divided by Total Exposure to Treatment |
| 3.5.1 | Number of Adverse Events, Serious Adverse Events, Fatal Adverse Events and Number of Adverse Events Causing Treatment Discontinuation |
| 3.5.2 | Number of Adverse Events by MedDRA System Organ Class |
| 3.5.3 | Number of Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.6 | Reasons for Seriousness for Serious Adverse Events |
| 3.7 | Serious Adverse Events |
| 3.7.1 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.7.2 | Number of Adverse Events by MedDRA System Organ Class and Preferred Term |

# **Psoriatic Arthritis**

| 1 | Baseline Characteristics- All Patients and Broken Down by Early Termination |
|---|---|
| 1.1 | Age |
| 1.2 | Gender |
| 1.3 | Disease Duration Before Inclusion |
| 1.4 | Anti-TNF use Before Inclusion |
| 1.4.1 | Anti-TNF Naïve / Experienced |
| 1.4.2 | Types of Anti-TNF use Before Inclusion |
| 1.5 | Physician's Assessment of Disease Activity |
| 1.6 | Clinical Examination |
| 1.6.1 | Joint Assessment (tender joints count, swollen joints count) |
| 1.6.2 | Inflammatory Parameters (CRP, ESR) |
| 1.6.3 | Physical Function (HAQ %) |
| 1.6.4 | BSA with Psoriasis |
| 1.6.5 | Patient's Numerical Rating Scale for Oligoarticular PsA Patients |
| 1.6.6 | Physician's Numerical Rating Scale for Oligoarticular PsA Patients |
| 1.7 | Concomitant Medication |
| 1.7.1 | Concomitant Steroids |
| 1.7.2 | Concomitant NSAIDs |
| 1.7.3 | Concomitant Immunomodulators |
| 1.7.4 | Number of DMARDs Used |
| 1.7.5 | Frequency of Use of Each Type of DMARD |
| 1.7.6 | Combination of Types of DMARD Used |
| 1.8 | Study Duration |
| 1.9 | Results of the Tests |
| 2 | Follow-up Data |
| <b>2</b> 2.1 | Follow-up Data Treatment Duration |
| | • |
| 2.1 | Treatment Duration |
| 2.1<br>2.1.1 | Treatment Duration Treatment Duration |
| 2.1<br>2.1.1<br>2.1.2 | Treatment Duration Treatment Duration Treatment Duration Category |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) in Each Window |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5<br>2.3.6 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) in Each Window Physical Function (HAQ %) - Difference from Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5<br>2.3.6 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) in Each Window Physical Function (HAQ %) - Difference from Baseline Physical Function (HAQ %) - Number of Patients with >7.33% Reduction from |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5<br>2.3.6<br>2.3.7 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) in Each Window Physical Function (HAQ %) - Difference from Baseline Physical Function (HAQ %) - Number of Patients with >7.33% Reduction from Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5<br>2.3.6<br>2.3.7 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) in Each Window Physical Function (HAQ %) - Difference from Baseline Physical Function (HAQ %) - Number of Patients with >7.33% Reduction from Baseline DAS28 in Each Window |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5<br>2.3.6<br>2.3.7 | Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) - Difference from Baseline Physical Function (HAQ %) - Number of Patients with >7.33% Reduction from Baseline DAS28 in Each Window DAS28 Category - Difference From Baseline |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.2<br>2.2.1<br>2.2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3<br>2.3.4<br>2.3.5<br>2.3.6<br>2.3.7<br>2.3.8<br>2.3.9<br>2.3.10 | Treatment Duration Treatment Duration Treatment Duration Category Treatment Duration Broken Down by Year of Start Treatment Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) Physician's Assessment of Disease Activity Physician's Assessment of Disease Activity in Each Window Physician's Assessment of Disease Activity - Difference from Baseline Clinical Examination Joint Assessment (tender joints count, swollen joints count) in Each Window Joint Assessment (tender joints count, swollen joints count) - Difference from Baseline Inflammatory Parameters (CRP, ESR) in Each Window Inflammatory Parameters (CRP, ESR) - Difference from Baseline Physical Function (HAQ %) in Each Window Physical Function (HAQ %) - Difference from Baseline Physical Function (HAQ %) - Number of Patients with >7.33% Reduction from Baseline DAS28 in Each Window DAS28 Category - Difference From Baseline DAS28 Category in Each Window |

- 2.3.14 Patient's Numerical Rating Scale for Oligoarticular PsA Patients Difference from Baseline
- 2.3.15 Physician's Numerical Rating Scale for Oligoarticular PsA Patients in Each Window
- 2.3.16 Physician's Numerical Rating Scale for Oligoarticular PsA Patients Difference from Baseline

#### **3** Adverse Events

- 3.1 Adverse Events
- 3.1.1 Patients with Adverse Events, Patients with Serious Adverse Events, Patients with Fatal Adverse Events and Patients with Adverse Events Causing Treatment Discontinuation
- 3.1.2 Patients with Adverse Events by MedDRA System Organ Class
- 3.1.3 Patients with Adverse Events by MedDRA System Organ Class and Preferred Term
- 3.2 Adverse Events per Year
- 3.2.1 Patients with Adverse Events, Patients with Serious Adverse Events, Patients with Fatal Adverse Events and Patients with Adverse Events Causing Treatment Discontinuation
- 3.2.2 Patients with Adverse Events by MedDRA System Organ Class
- 3.2.3 Patients with Adverse Events by MedDRA System Organ Class and Preferred Term
- 3.3 Adverse Events by Cumulative Yearly Period
- 3.3.1 Patients with Adverse Events, Patients with Serious Adverse Events, Patients with Fatal Adverse Events and Patients with Adverse Events Causing Treatment Discontinuation
- 3.3.2 Patients with Adverse Events by MedDRA System Organ Class
- 3.3.3 Patients with Adverse Events by MedDRA System Organ Class and Preferred Term
- 3.4 Incidence Adverse Events
- 3.4.1 Number of Adverse Events, Serious Adverse Events, Fatal Adverse Events and Number of Adverse Events Causing Treatment Discontinuation
- 3.4.2 Number of Adverse Events by MedDRA System Organ Class
- 3.4.3 Number of Adverse Events by MedDRA System Organ Class and Preferred Term
- 3.5 Incidence Adverse Events Divided by Total Exposure to Treatment
- 3.5.1 Number of Adverse Events, Serious Adverse Events, Fatal Adverse Events and Number of Adverse Events Causing Treatment Discontinuation
- 3.5.2 Number of Adverse Events by MedDRA System Organ Class
- 3.5.3 Number of Adverse Events by MedDRA System Organ Class and Preferred Term
- 3.6 Reasons for Seriousness for Serious Adverse Events
- 3.7 Serious Adverse Events
- 3.7.1 Patients with Adverse Events by MedDRA System Organ Class and Preferred Term
- 3.7.2 Number of Adverse Events by MedDRA System Organ Class and Preferred Term

# **Ankylosing Spondylitis**

| 1 | Baseline Characteristics- All Patients and Broken Down by Early Termination |
|---|---|
| 1.1 | Age |
| 1.2 | Gender |
| 1.3 | Disease Duration Before Inclusion |
| 1.4 | Anti-TNF use Before Inclusion |
| 1.4.1 | Anti-TNF Naïve / Experienced |
| 1.4.2 | Types of Anti-TNF use Before Inclusion |
| 1.5 | Physician's Assessment of Disease Activity |
| 1.6 | Clinical Examination |
| 1.6.1 | Joint Assessment (tender joints count, swollen joints count) |
| 1.6.2 | Inflammatory Parameters (CRP, ESR) |
| 1.6.3 | Physical Function (HAQ %) |
| 1.6.4 | Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) |
| 1.7 | Concomitant Medication |
| 1.7.1 | Concomitant Steroids |
| 1.7.2 | Concomitant NSAIDs |
| 1.7.3 | Concomitant Immunomodulators |
| 1.7.4 | Number of DMARDs Used |
| 1.7.5 | Frequency of Use of Each Type of DMARD |
| 1.7.6 | Combination of Types of DMARD Used |
| 1.8 | Study Duration |
| 1.9 | Results of the Tests |
| 2 | Follow-up Data |
| 2.1 | Treatment Duration |
| 2.1.1 | Treatment Duration |
| 2.1.2 | Treatment Duration Category |
| 2.1.3 | Treatment Duration Broken Down by Year of Start Treatment |
| 2.1.4 | Treatment Duration Broken Down by DAS28 Category at Window 2 (Month 6) |
| 2.2 | Physician's Assessment of Disease Activity |
| 2.2.1 | Physician's Assessment of Disease Activity in Each Window |
| 2.2.2 | Physician's Assessment of Disease Activity - Difference from Baseline |
| 2.3 | Clinical Examination |
| 2.3.1 | Joint Assessment (tender joints count, swollen joints count) in Each Window |
| 2.3.2 | Joint Assessment (tender joints count, swollen joints count) – Difference from |
| 2.3.2 | Baseline |
| 2.3.3 | Inflammatory Parameters (CRP, ESR) in Each Window |
| 2.3.4 | Inflammatory Parameters (CRP, ESR) – Difference from Baseline |
| 2.3.5 | Physical Function (HAQ %) in Each Window |
| 2.3.6 | Physical Function (HAQ %) – Difference from Baseline |
| 2.3.7 | Physical Function (HAQ %) - Number of Patients with >7.33% Reduction from |
| 2.3.7 | Baseline |
| 2.3.8 | DAS28 in Each Window |
| 2.3.9 | DAS28 Category – Difference From Baseline |
| 2.3.10 | DAS28 Category in Each Window |
| 2.3.10 | Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in Each Window |
| 2.3.11 | Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in Each window Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) - Difference from |
| 2.3.12 | Baseline Baseline |
| | Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) - Responder |

| 3 | Adverse Events |
|---|---|
| 3.1 | Adverse Events |
| 3.1.1 | Patients with Adverse Events, Patients with Serious Adverse Events, Patients with |
| | Fatal Adverse Events and Patients with Adverse Events Causing Treatment |
| | Discontinuation |
| 3.1.2 | Patients with Adverse Events by MedDRA System Organ Class |
| 3.1.3 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.2 | Adverse Events per Year |
| 3.2.1 | Patients with Adverse Events, Patients with Serious Adverse Events, Patients with |
| | Fatal Adverse Events and Patients with Adverse Events Causing Treatment |
| | Discontinuation |
| 3.2.2 | Patients with Adverse Events by MedDRA System Organ Class |
| 3.2.3 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.3 | Adverse Events by Cumulative Yearly Period |
| 3.3.1 | Patients with Adverse Events, Patients with Serious Adverse Events, Patients with |
| | Fatal Adverse Events and Patients with Adverse Events Causing Treatment |
| | Discontinuation |
| 3.3.2 | Patients with Adverse Events by MedDRA System Organ Class |
| 3.3.3 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.4 | Incidence Adverse Events |
| 3.4.1 | Number of Adverse Events, Serious Adverse Events, Fatal Adverse Events and |
| | Number of Adverse Events Causing Treatment Discontinuation |
| 3.4.2 | Number of Adverse Events by MedDRA System Organ Class |
| 3.4.3 | Number of Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.5 | Incidence Adverse Events Divided by Total Exposure to Treatment |
| 3.5.1 | Number of Adverse Events, Serious Adverse Events, Fatal Adverse Events and |
| | Number of Adverse Events Causing Treatment Discontinuation |
| 3.5.2 | Number of Adverse Events by MedDRA System Organ Class |
| 3.5.3 | Number of Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.6 | Reasons for Seriousness for Serious Adverse Events |
| 3.7 | Serious Adverse Events |
| 3.7.1 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.7.2 | Number of Adverse Events by MedDRA System Organ Class and Preferred Term |

# **All Patients**

| 3 | Adverse Events |
|---|---|
| 3.1 | Adverse Events |
| 3.1.1 | Patients with Adverse Events, Patients with Serious Adverse Events, Patients with Fatal Adverse Events and Patients with Adverse Events Causing Treatment Discontinuation |
| 3.1.2 | Patients with Adverse Events by MedDRA System Organ Class |
| 3.1.3 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.2 | Adverse Events per Year |
| 3.2.1 | Patients with Adverse Events, Patients with Serious Adverse Events, Patients with Fatal Adverse Events and Patients with Adverse Events Causing Treatment Discontinuation |
| 3.2.2 | Patients with Adverse Events by MedDRA System Organ Class |
| 3.2.3 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.3 | Adverse Events by Cumulative Yearly Period |
| 3.3.1 | Patients with Adverse Events, Patients with Serious Adverse Events, Patients with Fatal Adverse Events and Patients with Adverse Events Causing Treatment Discontinuation |
| 3.3.2 | Patients with Adverse Events by MedDRA System Organ Class |
| 3.3.3 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.4 | Incidence Adverse Events |
| 3.4.1 | Number of Adverse Events, Serious Adverse Events, Fatal Adverse Events and |
| J.T.1 | Number of Adverse Events, Serious Adverse Events, Fatar Adverse Events and Number of Adverse Events Causing Treatment Discontinuation |
| 3.4.2 | Number of Adverse Events by MedDRA System Organ Class |
| 3.4.3 | Number of Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.5 | Incidence Adverse Events Divided by Total Exposure to Treatment |
| 3.5.1 | Number of Adverse Events, Serious Adverse Events, Fatal Adverse Events and |
| | Number of Adverse Events Causing Treatment Discontinuation |
| 3.5.2 | Number of Adverse Events by MedDRA System Organ Class |
| 3.5.3 | Number of Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.6 | Reasons for Seriousness for Serious Adverse Events |
| 3.7 | Serious Adverse Events |
| 3.7.1 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.7.2 | Number of Adverse Events by MedDRA System Organ Class and Preferred Term |
| 3.8 | Non-Serious Adverse Events |
| 3.8.1 | Patients with Adverse Events by MedDRA System Organ Class and Preferred Term |